CLINICAL TRIAL: NCT05078034
Title: High-flow Nasal Oxygen With or Without Helmet Non-invasive Ventilation for Oxygenation Support in Acute Respiratory Failure (the HONOUR Pilot Trial)
Brief Title: HNFO With or Without Helmet NIV for Oxygenation Support in Acute Respiratory Failure Pilot RCT
Acronym: HONOUR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HONOUR (3693)
Record Dates: First submitted 2021-10-01; First posted 2021-10-14 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-04

CONDITIONS: Acute Hypoxemic Respiratory Failure
Keywords: High Flow Nasal Oxygen; Helmet Non Invasive Ventilation
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: 1:1 randomized control trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HFNO (Active Comparator): High Flow Nasal Oxygen alone
  Interventions: Device: High Flow Nasal Oxygen
- H-NIV (Active Comparator): Helmet Non-Invasive ventilation for a minimum of 12 hours per day with HFNO between sessions
  Interventions: Device: Helmet Non-Invasive Ventilation (HNIV)

INTERVENTIONS:
Device: Helmet Non-Invasive Ventilation (HNIV) — HNIV will be connected to a ventilator by a conventional closed respiratory circuit. Sessions of HNIV will be delivered with PEEP targeting a minimum 12 hours/day. PEEP will be titrated according to patient comfort, work of breathing, and O2 saturation. Pressure support will be titrated to lowest level tolerated. Between HNIV sessions, patients will be supported with HFNO at the same required FiO2. Starting on study day 3, patients will be screened for discontinuation of HNIV. Once HNIV is stopped, patients will be transitioned to HFNO and then weaned from HFNO as tolerated.
  Other Names: HNIV
  Arms: H-NIV
Device: High Flow Nasal Oxygen — HFNO will be provided. FiO2 will be titrated to achieve a target O2 saturation of 92-97%, and flows will be initiated at 50 litres/minute and titrated as per usual practice for comfort and oxygenation. Once the target O2 saturation is achieved, the FiO2 will be titrated to the minimal value to maintain this target saturation. HFNO will be provided continuously over a minimum of 2 calendar days. Starting on study day 3, patients will be weaned from HFNO as tolerated.
  Other Names: HFNO
  Arms: HFNO

SUMMARY:
This Randomized Control Trial will directly compare helmet non-invasive ventilation (NIV) combined with high flow nasal oxygen (HFNO) versus HFNO alone in patients with Acute Hypoxemic Respiratory Failure (AHRF).

DETAILED DESCRIPTION:
This is a pilot multicentre, concealed, stratified, permuted block randomized controlled trial enrolling patients with AHRF who are admitted to the intensive care unit. Patients with imminent need for intubation, or a contraindication to study interventions will be excluded. Patients will be randomized to receive either (1) sessions of at least 12 hours per day of helmet NIV oxygen interspersed with HFNO or (2) HFNO alone over at least 2 calendar days. Participants will be followed to hospital discharge or 60 days, with an additional quality of life assessment via telephone interview 6 months after enrolment.

ELIGIBILITY:
Inclusion Criteria:

1. Intensive care unit admission (orders written)
2. Age ≥18 years
3. Hypoxemic acute respiratory failure for at least 1 hour and still present at time of screening for eligibility (symptom onset during last 14 days) with the following:

   1. Respiratory rate >21bpm or clinical evidence of increased work of breathing and
   2. Documented Hypoxemia defined as any one of:

   i. PaO2:FiO2 < 300 ii. If no arterial blood gas available, then SpO2:FiO2 < 315 iii. Oxygen saturation <98% on FiO2 >= 0.4 or higher by Venturi mask, TAVISH mask 10 Litres / minute, or any non-invasive oxygenation strategy
4. Not already intubated or with tracheostomy

Exclusion Criteria:

1. Already on HFNO or other non-invasive ventilation strategy at FiO2>=0.4 for the last 24 hours in the ICU.
2. Immediate need for intubation (e.g., inadequate airway protection or refractory hypoxemia or cardiopulmonary arrest, massive hemoptysis, etc)
3. Extubated in the ICU within past 72 hours
4. Clinician deems that face mask NIV is indicated to treat a primary diagnosis of hypercapnic respiratory failure or acute congestive heart failure
5. Known neuromuscular disease
6. Patients being transitioned to Palliative care or unlikely to survive more than 24 hours
7. ICU discharge is planned or anticipated on the day of screening
8. Previously enrolled in this trial
9. Trauma patients who remain in a cervical spine collar at the time of recruitment or who have upper limb/torso fractures that would preclude them from safe application of the helmet
10. Clinician decision that positive pressure to face and/or nasal pharynx is a contraindication (eg. Transphenoidal surgery, basal skull fracture etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-03-17 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rates | 2 years
  Recruitment rate at different study sites
Non-randomized Eligible Patients | 2 years
  Proportion of Eligible patients who are not randomized and reasons for this
Adherence/Compliance to Oxygenation Strategy | 2 years
  Rate of adherence to the assigned oxygenation strategy (and crossover rates)
Among patients requiring intubation in each group, the number who were intubated according to the pre-specified criteria | 2 years
  Adherence to pre-specified criteria for intubation in each group
Time from ICU admission to randomization and initiation of treatment | 2 years
  Median time from ICU admission to randomization and initiation of the allocated treatment

SECONDARY OUTCOMES:
Number of participants in each group who need endotracheal intubation | 28 and 60 days
  Need for endotracheal intubation after randomization
Duration of invasive mechanical ventilation after randomization up to 28 and 60 days | 28 and 60 days
  Duration of invasive mechanical ventilation after randomization up to 28 and 60 days
Duration of non-invasive respiratory support after randomization up to 28 and 60 days | 60 days
  Duration of non-invasive mechanical ventilation after randomization up to 60 days
ICU length of stay | 28 days
  days of ICU up to 28 days after randomization
All cause mortality | 60 days
  All cause mortality to 60 days
COVID-19 infection after hospitalization | 28 days
  diagnosis of COVID-19
Health related quality of life | 180 days
  Health related quality of life as measured by telephone using the European Quality of Life Five Dimension (EQ-5D) tool, where a score of 1 means the patient has no problems, and a score of 5 mean the patient has extreme problems in the 5 dimensions.
Mortality at 180 days | 180 days
  Mortality to 180 days
Activities of Daily Living | 180 days
  Katz Index of Independence in Activities of Daily Living (ADL) where a high of 6 means the patient can perform the activities fully independently, and a low of 0 means the patient is fully dependent and unable to perform activities without assistance.
Ventilator-Free Days to day 28, analyzed as an ordinal variable, with death = 0 days | 28 days
  Ventilator-Free Days to day 28, analyzed as an ordinal variable, with death = 0 days

CONTACTS AND LOCATIONS:
Overall Officials: Damon Scales, MD PhD FRCPC, Principal Investigator — Sunnybrook Health Sciences Centre; Niall Fergusson, MD FRCPC, Principal Investigator — University Health Network, Toronto
Locations (11):
- Canada (11):
  - University of Calgary, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Hamilton Health Sciences- Juravinski, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - London Health Sciences Centre, London, Ontario
  - Ottawa Hospital, Ottawa, Ontario
  - North York General Hospital, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - University Health Network Toronto General, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Angriman F, Ferreyro BL, Rochwerg B, Sklar M, Adhikari N, Bagshaw SM, Brochard L, Cuthbertson B, Del Sorbo L, Fowler R, Geagea A, Granton JT, Mehta S, Munshi L, Muscedere J, Nardi J, Parhar K, Pinto RL, Piquette D, Seely A, Slessarev M, Tobin S, Scales DC, Ferguson ND; HONOUR Investigators and the Canadian Critical Care Trials Group. High-flow nasal Oxygen with or without alternating helmet Non-invasive ventilation for Oxygenation sUpport in acute Respiratory failure (HONOUR): a protocol for a pilot randomised controlled trial. BMJ Open. 2025 Oct 27;15(10):e111526. doi: 10.1136/bmjopen-2025-111526. PMID 41145249